CLINICAL TRIAL: NCT02369250
Title: Rosuvastatin 1.2mg in Situ Gel Combined With 1:1 Mixture of Autologous Platelet-rich Fibrin and Porus- Hydroxyappatite Bone Graft in Surgical Treatment of Mandibular Degree II Furcation Defects: A Randomized Clinical Control Trial
Brief Title: Rosuvastatin Gel With 1:1 Mixture of Platelet-rich Fibrin and Bone Graft in Mandibular Degree II Furcation Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Proffesor and Head, dept of periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/12/2013-14
Record Dates: First submitted 2014-12-04; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Furcation Defects
Keywords: regeneration; surgical therapy; furcation defect
MeSH Terms: conditions — Furcation Defects | interventions — Rosuvastatin Calcium; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OFD+ PLACEBO GEL (Placebo Comparator): furcation defect site is surgically debrid and placed a placebo gel
- OFD+ PRF + BONE GRAFT (Active Comparator): Following surgical debridment of furcation site autologous PRF and bone graft is placed in defect as a competator drug used is platelet rich fibrin and porus hydroxyapatite bone graft
  Interventions: Biological: platelet rich fibrin
- RSV1.2% gel + PRF+ BG (Experimental): Following surgical debridment of furcation site Rosuvastatin 1.2% in situ gel combined with autologous PRF and bone graft is placed
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin, is a statin group of drug.
  Other Names: statin
  Arms: RSV1.2% gel + PRF+ BG
Biological: platelet rich fibrin — AUTOLOGUS PLATELET GROWTH FACTOR
  Other Names: platelet concentrate
  Arms: OFD+ PRF + BONE GRAFT

SUMMARY:
Rosuvastatin (RSV) is a new synthetic, second-generation, sulfur-containing, hydrophilic statin, that stimulate bone formation in critical-size cortical bone defects adjacent to titanium implants, when administered locally in bone. Platelet-rich fibrin (PRF) is a platelet concentrate with sustained release of various growth factors, having regenerative potential to treat periodontal defects. Porous hydroxyapatite (HA) bone grafting material has clinically satisfactory response, when used to fill periodontal intrabony defects. This double-masked randomized study is designed to evaluate the potency of combination of RSV 1.2mg in situ gel with 1:1 mixture of autologous PRF and HA bone graft in the surgical treatment of mandibular degree II furcation defects when compared with autologous PRF and HA bone graft placed after open flap debridement (OFD).

DETAILED DESCRIPTION:
ABSTRACT Background: A wide range of regenerative materials have been tried in the treatment of furcation defects. Rosuvastatin (RSV) is a new synthetic, second-generation, sulfur-containing, hydrophilic statin, that stimulate bone formation in critical-size cortical bone defects adjacent to titanium implants, when administered locally in bone. Platelet-rich fibrin (PRF) is a platelet concentrate with sustained release of various growth factors, having regenerative potential to treat periodontal defects. Porous hydroxyapatite (HA) bone grafting material has clinically satisfactory response, when used to fill periodontal intrabony defects. This double-masked randomized study is designed to evaluate the potency of combination of RSV 1.2mg in situ gel with 1:1 mixture of autologous PRF and HA bone graft in the surgical treatment of mandibular degree II furcation defects when compared with autologous PRF and HA bone graft placed after open flap debridement (OFD).

Material and methods 105 patients with mandibular buccal Class II furcation defects were randomly allotted and treated either with, OFD and placebo gel: Group 1, or OFD + autologous PRF and porus-HA bone graft: Group 2, or OFD + RSV 1.2mg in situ gel combined with autologous PRF and porus-HA bone graft: Group 3. Clinical parameters were recorded at baseline before SRP and at 9 months; they included modified sulcus bleeding index (mSBI), probing depth (PD), and relative vertical (RVAL) and horizontal (RHAL) attachment levels. At baseline and after 9 months, radiographic assessment of bone defect fill was performed postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. the presence of buccal Class II furcation defects in endodontically vital, asymptomatic mandibular first and second molars with a radiolucency in the furcation area on an intraoral periapical radiograph with PD ± 5mm and horizontal PD ± 3mm after Phase I therapy (SRP)
2. no history of antibiotic or periodontal therapy in the preceding 6 months.

Exclusion Criteria:

1. systemic illness known to affect the outcomes of periodontal therapy, such as diabetes mellitus, cardiac diseases, insufficient platelet count (<200,000/mm3), or immunocompromised (e.g., HIV individuals) patients taking medications, such as corticosteroids or calcium channel blockers, which are known to interfere with periodontal wound healing
2. individuals known or suspected allergy to the RSV group or allergic to medications
3. systemic statin therapy
4. pregnant or lactating women
5. patients using tobacco in any form
6. individuals with unacceptable oral hygiene (plaque index >1.5). In addition, teeth with interproximal intrabony defects, gingival recession, endodontic (pulpal) involvement, or mobility of tooth ≥ Grade II were also excluded.

Ages: 26 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
BONE FILL | 9 MONTHS
  BONE FILL/ defect depth reduction recorded at baseline and at 9 months

SECONDARY OUTCOMES:
Probing depth | 9 months
  Probing depth recorded at baselin and at 9 months
Clinical attachment level | 9 months
  Gain in Clinical attachment level from cementoenamel junction to the base of the periodontal pocket